CLINICAL TRIAL: NCT04229524
Title: Quantitative Assessment of the Correlation Between Blood Supply in the Gastic Conduit and the Incidence of Anastomotic Fistula With Fluorescence Angiography for Esophageal Reconstruction
Brief Title: Quantitative Assessment of Blood Supply in the Gastic Conduit With Fluorescence Angiography for Esophageal Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yongtao Han, Director,Head of Thoracic Surgery, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2001
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; blood supply; anastomotic fistula; fluorescence angiography
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- angiographic intervention group (Experimental): Enrolled patients will undergo thoracoscopy combined with a three-incision esophageal carcinoma radical mastectomy and two-field (chest-abdomen) lymph node dissection.Quantitative assessment of blood supply in the gastic conduit was performed using fluoroscopy before esophagogastric anastomosis.
  Interventions: Procedure: Fluorescence angiography
- control group (No Intervention): The same surgical method as the experimental group.The only difference is that the position of the gastic conduit anastomosis is determined based on the experience of the doctor.

INTERVENTIONS:
Procedure: Fluorescence angiography — After the tube and stomach were made during surgery, the predetermined anastomosis position was marked with sutures in advance according to the doctor's experience, and then 0.04ml / kg indocyanine green injection was injected into the central vein. Next, dynamic observation and recording of the tube-gastric anastomosis area in 136 seconds using a fluorescent imaging system with a fixed focal length till the fluorescence reaching range and intensity. If the average value of the fluorescence value of the anastomosis position is greater than 30, then the anastomosis position may be according to the original plan or moved to the proximal part. If the average fluorescence value of the predetermined anastomosis position is less than 30, the anastomosis must move to proximal part ensure anastomosis with fluorescence value at least> 30.
  Arms: angiographic intervention group

SUMMARY:
A single-institution, randomize controlled trial is to be held to evaluate the correlation between blood supply in the gastic conduit and the incidence of anastomotic fistula during radical operation for esophageal squamous cell carcinoma by fluorescence angiography.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically confirmed esophageal squamous cell carcinoma and and potential resection;
* 2.Intend to undergo thoracic laparoscopy combined with three-incision esophageal cancer radical operation;
* 3.The stomach is used as an esophageal substitute for reconstruction;
* 4.Enrolled patients will adopt the esophagus bed pathway and round neck anastomosis method;
* 5.Have a performance status of 0 or 1 on the ECOG Performance Scale; Adequate organ function;
* 6.Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

* 1.Histologically confirmed non-squamous cell carcinoma of the esophagus ;
* 2.The ECOG score of patient's physics >1;
* 3.Patients who use other organs instead of the esophagus;
* 4.Patients with vascular arch injury and need vascular anastomosis;
* 5.Patients with multiple complications such as heart disease or diabetes;
* 6.Other patients whom the medical practitioner considers inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of anastomotic fistula | 3 months
  Anastomotic fistula is defined as an anastomotic fistula or any anastomotic dehiscence or leakage of saliva from a neck wound, confirmed by gastroscopy or upper gastrointestinal angiography, or purulent discharge from the chest or mediastinal drainage catheter. In addition, in this study, occult fistula was not included in the anastomotic fistula group when invasive treatment was not required.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

REFERENCES:
- [Derived] He W, Li Z, Deng X, Zheng K, Wang C, Peng L, Han Y, Leng X, Zhou Q. Fluorescence quantitative assessment of blood perfusion in the gastric conduit to reduce anastomotic leakage after esophagectomy: a randomized controlled trial. Surg Endosc. 2025 Oct;39(10):6644-6654. doi: 10.1007/s00464-025-12093-6. Epub 2025 Aug 20. PMID 40835759